

## Information and Consent page for an Online Survey/Questionnaire

Study Title: The impact of a bespoke mindfulness intervention for Registered Dietitians. A randomised controlled trial.

#### **Research Team:**

Dr. Amanda Avery (Principal Investigator, PhD Supervisor), School of Biosciences, University of Nottingham

Lynsey Richards (PhD Student), School of Biosciences, University of Nottingham

Jake Sallaway-Costello (PhD Co-Supervisor), School of Biosciences, University of Nottingham

## Faculty of Medicine & Health Sciences Research Ethics Ref: FMHS XXXX

The aim of this study is to determine the impact of a bespoke mindfulness education package (the intervention) compared with a control group (a group of Registered Dietitians who do not receive the intervention). We would also like to find out about the barriers and facilitators to incorporating mindfulness into dietetic practice.

You are invited to participate in this research study if you are:

- A Registered Dietitian currently practicing in the UK
- Willing and able to participate in 4 x 50 minute CPD sessions relating to mindfulness in dietetic practice (one session per week)
- Willing and able to complete all of the surveys (pre-intervention, immediately post, 3 months post and 6 months post intervention)

Please read through this information before agreeing to participate. You can ask any questions before deciding by contacting the researchers (details below). Taking part is entirely voluntary.

### What will I be asked to do?

The first phase of this research will involve measuring levels of resilience, stress and burnout using pre-existing, validated questionnaires before the intervention. This will be in the form of an online survey and will take around 20 minutes to complete. The survey is anonymous. This survey will be repeated immediately after, 3 months after and 6 months after the intervention. All participants will be asked to complete the surveys.

Following completion of the pre-intervention survey, all participants will be randomly allocated to either the intervention or the control group. Those allocated to the intervention group will be invited to participate in the mindfulness CPD (4 x 50 minute online mindfulness sessions). Those allocated to the control group (waitlist) will not receive the intervention initially, but will still be sent the surveys at the intervals specified above. Following the completion of the study, the waitlist group will all be offered the same CPD as the intervention group. No further surveys or interviews will be requested after that point.



The second phase of this research will be a one off, individual interview, conducted 6 months after the intervention, exploring the experiences of the participant in relation to incorporating mindfulness practice into their working life. Interviews will take around 30 – 45 minutes, will be hosted online and will be audio recorded, then transcribed. All audio recordings will be deleted following transcription. All transcripts will be anonymised. You can indicate at the end of this page whether or not you want to be contacted to be interviewed. Whether or not you would like to be considered for interview will not affect your participation in the first phase of the study. If you do wish to be considered for interview, you will be sent further information closer to the time and will be free to either accept or decline the invitation.

# What are the disadvantages of taking part?

Participating in the research *may* involve recalling stressful or difficult experiences but is not anticipated to cause you significant disadvantages or discomfort. The potential psychological harm or distress should not exceed that experienced in everyday life.

# What are the advantages of taking part?

All participants in this study will have access to a free, bespoke mindfulness CPD, developed especially for Registered Dietitians.

By taking part in the intervention and engaging in the data collection (interviews and / or surveys), you will be contributing data to a topic that lacks robust research and where dietitians are underrepresented as a professional group.

# Will my answers be kept confidential?

All responses to the survey are anonymous. Interview transcripts will be anonymised. All information collected during the course of the research will be kept strictly confidential. You will not be able to be identified in any reports or publications. Data collected in the online questionnaire will be stored online in a form protected by passwords and other relevant security processes and technologies. Data collected may be shared in an anonymised form to allow reuse by the research team. These anonymised data will not allow any individuals or their institutions to be identified or identifiable.

# What if I decide I no longer wish to take part?

During the course of the study, a participant may choose to withdraw at any time. This may happen for several reasons, including but not limited to:

- Distress during survey completion, intervention or interview
- Inability to comply with study procedures
- Participant decision

When completing the surveys, you will be prompted to enter a code (the last 3 digits of your phone number and the last 3 digits of your postcode) in order to allow us to match your responses throughout the study, but also to allow us to identify your responses should you wish to withdraw your data at a later time.



If you decide to withdraw, but have already completed a survey or interview, you can either leave your data in the dataset and not engage further with the study, or you can request that your survey responses and / or transcript is deleted, up until 1st February 2025 after which point, your data will have been processed for analysis and it will no longer be possible to remove your data from the dataset.

In addition, the investigator may discontinue your participation due to ineligibility (either arising during the study or retrospectively being overlooked or not disclosed at screening. This will result in exclusion of your data from analysis, if possible.

## What will happen to your data?

All anonymised research data created by the project will be stored in a password protected folder within a restricted access server at the University of Nottingham. In addition, anonymised data will be deposited to the research data archive. University of Nottingham will retain and preserve research data in line with University requirements for a minimum of 7 years, but data will be retained for longer periods of time where it is of continual value to users.

This intervention and the associated surveys are part of a PhD thesis. The results will be written up as a research project and may be used in academic publications and presentations. The overall anonymised data from this study may be shared for use in future research and teaching (with research ethics approval). It will not be possible to identify you from any publications or presentations.

The only personal data we will receive is your e-mail when you register your interest to participate. This will be received and handled separately from your completed questionnaire and it will not be possible to link the sets of data. Your e-mail address will only be kept as long as needed to invite you to the intervention and to send you survey links. It will then be destroyed. For further information about how the university processes personal data please see:

https://www.nottingham.ac.uk/utilities/privacy.aspx/

### Who will have access to your data?

The University of Nottingham is the data controller (legally responsible for data security) and the Supervisor of this study (named above) is the data custodian (manages access to the data) and as such will determine how your data is used in the study. Your research and personal data will be used for the purposes of the research only. Research is a task that we perform in the public interest.

Responsible members of the University of Nottingham may be given access to data for monitoring and/or audit of the study to ensure it is being carried out correctly.

If you have any questions or concerns about this project, please contact:

Lynsey Richards E-mail: <a href="mailto:lynsey.richards@nottingham.ac.uk">lynsey.richards@nottingham.ac.uk</a>

or if you have any concerns about any aspect of this study please contact the Principal Investigator: Dr Amanda Avery E-mail: <a href="mailto:Amanda.Avery@nottingham.ac.uk">Amanda.Avery@nottingham.ac.uk</a>).



If you remain unhappy and wish to complain formally, you should then contact the FMHS Research Ethics Committee Administrator E-mail: <a href="mailto:FMHS-ResearchEthics@nottingham.ac.uk">FMHS-ResearchEthics@nottingham.ac.uk</a>

If you would like to discuss the research with someone beforehand (or if you have questions afterwards), please contact:

Lynsey Richards
PhD Student - School of Biosciences

Email: <a href="mailto:lynsey.richards@nottingham.ac.uk">lynsey.richards@nottingham.ac.uk</a>

**Consent** (Only if the respondent provides consent by choosing "I confirm all of the above statements are true and give consent to participate in this study" from a drop down will they be able to access the survey questions. The other option is "I do not consent / I do not meet the criteria set out above", which will skip the respondent straight to the end page, without offering them the survey questions)

### I confirm that:

I have read and understood the participant information sheet

I have had the opportunity to ask questions

I understand that participation for any stage of the study is entirely voluntary

I understand that I have the right to withdraw at any stage of the study without prejudice

I understand my right to anonymity and confidentiality

I am a HCPC Registered Dietitian, currently practicing in the UK

I do not have a diagnosis of a psychotic condition

I do not have a diagnosis of epilepsy or asthma OR I have well controlled asthma or epilepsy OR I have been given permission from an appropriate medical doctor to participate in this intervention